CLINICAL TRIAL: NCT02184039
Title: Clinical Therapeutic Evaluation Program in Patients With Rheumatic Diseases
Brief Title: Efficacy and Safety of Meloxicam (Mobicox®) in Mexican Population With Rheumatic Diseases
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 107.264
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Study to evaluate the efficacy and safety of meloxicam (Mobicox®) in Mexican population with rheumatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* none

Exclusion Criteria:

* Hypersensitivity to meloxicam or to other NSAIDS
* History of asthma, angioedema or urticaria secondary to NSAIDS
* Pregnancy or lactation
* Recent or current history of peptic ulcer disease, severe renal failure, severe hepatic failure
* Age below of 12 years.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 12687 (Actual)
Dates: Start 2003-05; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Change in intensity of the symptoms measured with a four-point scale | Baseline, 30 and 90 days

SECONDARY OUTCOMES:
Degree of satisfaction evaluated with a six point numerical rating scale | up to 90 days
Number of patients with adverse events | up to 90 days